CLINICAL TRIAL: NCT06116981
Title: Effects of High-induction Magnetic Field Therapy in Patients With Shoulder Pain
Brief Title: High-induction Magnetic Field Therapy in Patients With Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KaratayU5
Record Dates: First submitted 2023-10-14; First posted 2023-11-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-10

CONDITIONS: Rehabilitation
Keywords: Magnetic Field Therapy; Shoulder Pain; Range of Motion
MeSH Terms: conditions — Shoulder Pain | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Group 1: Conservative Treatment Group Grou 2: Conservative Treatment + High Induction Magnetic Field Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group consists of individuals who received high-induction magnetic field therapy in addition to conservative treatment (routine rehabilitation sessions including stretching, transcutaneous electrical nerve stimulation, and exercises.).
  Interventions: Other: High Induction Magnetic Field Therapy; Other: Conservative Treatment
- Comparison Group (Active Comparator): Conservative Treatment Group: Group with routine rehabilitation sessions including stretching, transcutaneous electrical nerve stimulation, and exercises.
  Interventions: Other: Conservative Treatment

INTERVENTIONS:
Other: High Induction Magnetic Field Therapy — High Induction Magnetic Field Therapy is a method that has no side effects, is non-invasive and easy to apply, and is used to increase circulation in tissues.
  Arms: Experimental Group
Other: Conservative Treatment — Shoulder exercises, transcutaneous electrical nerve stimulation, stretching.

SUMMARY:
High Induction Magnetic Field Therapy is a therapeutic method that uses high-intensity fields (up to 2.5 T) that produce high current density in exposed tissue. While there are studies in the literature on devices with 2.5 T, there is no research on the effect of 4 T. Magnetic field application contributes significantly to the healing process. It is an easier, cheaper, and more comfortable application. The magnetic field has been clinically proven to be safe. It is a practical, non-invasive method to induce cell and tissue modifications, correcting selected pathological conditions through magnetic application. The aim of the study is to investigate whether High Induction Magnetic Field therapy applied in addition to conservative treatment in patients with shoulder pain makes a difference compared to conservative treatment alone.

DETAILED DESCRIPTION:
It is planned to include people between the ages of 18-65 in the study. Before the evaluation, written consent will be obtained from the participants and information on their age, gender, weight, height, chronic disease and medication use, presence of previous surgical operations, daily activity frequency, alcohol or cigarette use will be obtained.

Individuals who voluntarily agree to participate in the study and have at least one of the following diagnoses: shoulder impingement syndrome, rotator cuff rupture, and subacromial bursitis will be included in the study. Individuals with a neurological, orthopedic or cardiovascular chronic disease that cannot be controlled with medication, those who are pregnant or suspected of being pregnant, those with a pacemaker, those with implanted ear hearing aids and those with metallic implants will be excluded.

Individuals' shoulder pain levels, normal joint range of motion and daily living activities will be evaluated before and after treatment.

It is planned to include two separate groups in the study: a conservative treatment group and a group that will receive high induction magnetic field therapy in addition to conservative treatment. Within the scope of conservative treatment, ice application, transcutaneous electrical stimulation-TENS, interferential current, stretching and strengthening exercises, and normal joint range of motion exercises will be applied. Conservative treatment will be continued five days a week for a total of four weeks. High induction magnetic field therapy (Salus Talent, 4 T) will be applied in 10 sessions, 10 minutes, with one day intervals within a four-week treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agreeing to participate in the research.
* Being between the ages of 18 and 65
* Having at least one of the following diagnoses: shoulder impingement syndrome, rotator cuff rupture, and subacromial bursitis.
* Having the cognitive fitness to perform the surveys and tests to be used during the research.

Exclusion Criteria

* Having a chronic disease such as neurological, orthopedic or cardiovascular that cannot be controlled with medication.
* Not volunteering to participate in the research.
* Pregnant and suspected pregnancy individuals
* Individuals with pacemakers
* Individuals with implantable ear hearing aids
* Individuals with metallic implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale-VAS | baseline and after 4 weeks of treatment
  A score between 0 and 10 points is given and used to evaluate pain.
Range of Motion | baseline and after 4 weeks of treatment
  Range of Motion of Shoulder Joint: Shoulder joint flexion (0-180 degrees), abduction (0-180 degrees), external rotation (0-90 degrees) and internal rotation (0-90 degrees) range of motion will be measured with a goniometer. Higher values indicate increased mobility.
Disabilities of the Arm, Shoulder and Hand (DASH) | baseline and after 4 weeks of treatment
  The DASH is a 30-item patient-reported outcome measure utilized to assess symptoms and function of the entire upper extremity. Total scores range from 0 (minimum) to (100) maximum. The first 30 questions of the survey will be applied. As the score increases, the disability level increases.
Constant Murley Score | baseline and after 4 weeks of treatment
  It is a 100-point scale consisting of 15 points for pain, 20 points for daily activities, 40 points for pain-free joint range of motion, and 25 points for strength parameters. While pain and daily living activities are evaluated by the patient, joint range of motion and strength are evaluated by the clinician. A higher score corresponds to a higher-quality of function.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Akkoyun Sert, PhD, Study Director — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No